CLINICAL TRIAL: NCT00584727
Title: Evaluation of Fit and Visual Acuity of the Cypress Toric Lens in Two Phases: Part A: A Non-Dispensing Comparison to SofLens66® Toric and Acuvue® 2
Brief Title: In-office Evaluation of Two Toric Soft Contact Lenses and a Spherical Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Foresight Regulatory Strategies, Inc. (Industry)
Responsible Party: Kurt Moody, OD, FAAO./ Manager, Clinical Research, Vistakon
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0714A
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Astigmatism
Keywords: astigmatism; visual acuity; fit; comfort; satisfaction; contact lens
MeSH Terms: conditions — Astigmatism; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- senofilcon A/alphafilcon A/etafilcon A (Active Comparator): First intervention:senofilcon A toric contact lenses Second intervention: alphafilcon A toric contact lenses Third intervention: etafilcon A sphere contact lenses
  Interventions: Device: senofilcon A toric contact lens; Device: alphafilcon A toric; Device: etafilcon A sphere
- alphafilcon A/etafilcon A/senofilcon A (Active Comparator): First intervention: alphafilcon A toric contact lenses Second intervention: etafilcon A sphere contact lenses Third intervention: senofilcon A toric contact lenses
  Interventions: Device: senofilcon A toric contact lens; Device: alphafilcon A toric; Device: etafilcon A sphere
- etafilcon A/senofilcon A/alphafilcon A (Active Comparator): First intervention: etafilcon A sphere contact lenses Second intervention:senofilcon A toric contact lenses Third intervention: alphafilcon A toric contact lenses
  Interventions: Device: senofilcon A toric contact lens; Device: alphafilcon A toric; Device: etafilcon A sphere
- senofilcon A/etafilcon A/alphafilcon A (Active Comparator): First intervention: senofilcon A toric contact lenses Second intervention: etafilcon A sphere contact lenses Third intervention: alphafilcon A toric contact lenses
  Interventions: Device: senofilcon A toric contact lens; Device: alphafilcon A toric; Device: etafilcon A sphere
- alphafilcon A/senofilcon A/etafilcon A (Active Comparator): First intervention: alphafilcon A toric contact lenses Second intervention: senofilcon A toric contact lenses Third intervention: etafilcon A sphere contact lenses
  Interventions: Device: senofilcon A toric contact lens; Device: alphafilcon A toric; Device: etafilcon A sphere
- etafilcon A/alphafilcon A/senofilcon A (Active Comparator): First intervention: etafilcon A sphere contact lenses Second intervention: alphafilcon A toric contact lenses Third intervention: senofilcon A toric contact lenses
  Interventions: Device: senofilcon A toric contact lens; Device: alphafilcon A toric; Device: etafilcon A sphere

INTERVENTIONS:
Device: senofilcon A toric contact lens — contact lens
Device: alphafilcon A toric — contact lens
Device: etafilcon A sphere — contact lens

SUMMARY:
The purpose of this study is to determine the relative performance of a new toric soft contact lens against a toric and a spherical contact lens currently available in market, specifically with regards to the fit and visual acuity as well as the comfort, vision and satisfaction while in the practitioner's office. Approximately 2 hours duration.

DETAILED DESCRIPTION:
Non-dispensing, single-masked (subject-masked), randomised, controlled study.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 and less than or equal to 39 years of age and have a need for vision correction in BOTH eyes (monovision or uniocular fitting is NOT allowed).
2. be of Asian descent (Japanese, Chinese, Korean, Polynesian or other Asian ancestry) and have Asian Eye anatomy
3. have successfully worn toric or spherical soft (hydrogel or silicone hydrogel) contact lenses for at least 4-weeks prior to enrollment in the study.
4. be able and willing to adhere to the instructions set forth in the protocol.
5. agree to wear their contact lenses in both eyes on a daily wear schedule for at least 8 hours per day every day during the study.
6. have a distance spherical component between -1.00 D and -5.50 D with cylinder in the range of 0.75 D to 2.25 D and cylinder axis within 10 ° of the vertical and within 20 ° of the horizontal in both eyes
7. have a best corrected manifest refraction visual acuity of at least 20/25 or better in each eye.
8. be in good general health, based on his/her knowledge.
9. read, be given an explanation of, indicate understanding of, and sign the STATEMENT OF INFORMED CONSENT.

Exclusion Criteria:

1. The subject is a rigid gas permeable (RGP) or daily disposable soft lens wearer.
2. The presence of clinically significant (grade 3 or 4) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids, or associated structures.
3. The presence of ocular or systemic disease or need for medication which might interfere with contact lens wear or which would cause the lenses to be removed more than twice a day. (i.e., Sjögren's syndrome, type II diabetes, etc).
4. Slit lamp findings that would contraindicate contact lens wear such as:

   * Pathological dry eye or associated findings
   * Pterygium or corneal scars within the visual axis
   * Neovascularization >1mm in from the limbus
   * History of giant papillary conjunctivitis (GPC) worse than Grade 2
   * Anterior uveitis or iritis (past or present)
   * Seborrhoeic eczema, seborrhoeic conjunctivitis
5. A history of recurrent erosions, corneal infiltrates, corneal ulcer or fungal infections.
6. A known history of corneal hypoesthesia (reduced corneal sensitivity.)
7. Aphakia, keratoconus or a highly irregular cornea.
8. Current pregnancy or lactation (to the best of the subject's knowledge).
9. Active participation in another clinical study at any time during this study.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chin, O.D., Principal Investigator; James Fujimoto, O.D., Principal Investigator; Weslie Hamada, OlD., Principal Investigator — Arthur T. Kobayashi, O.D., Inc.; Dennis Kuwuabara, O.D., Principal Investigator — Eye Care Associates of Hawaii; Mark Nakano, O.D., Principal Investigator — Mark E. Nakano Optometric Corp.; Ikuko Sugimoto, O.D., Principal Investigator; Kevin Rosin, O.D., Principal Investigator — Drs. Farkas, Kassalow, Resnick & Associates; Jennifer Kao, O.D., Principal Investigator

RESULTS

PARTICIPANT FLOW:
Groups:
- Senofilcon A/Alphafilcon A/Etafilcon A: First Intervention: senofilcon A toric contact lenses Second Intervention: alphafilcon A toric contact lenses Third Intervention: etafilcon A sphere contact lenses
- Etafilcon A/Senofilcon A/Alphafilcon A: First Intervention: etafilcon A sphere contact lenses Second Intervention: senofilcon A toric contact lenses Third Intervention: alphafilcon A toric contact lenses
- Alphafilcon A/Senofilcon A/Etafilcon A: First intervention: alphafilcon A toric Second intervention: senofilcon A toric Third intervention: etafilcon A sphere
Period: First Intervention
Arm/Group | Senofilcon A/Alphafilcon A/Etafilcon A | Alphafilcon A/Etafilcon A/Senofilcon A | Etafilcon A/Senofilcon A/Alphafilcon A | Senofilcon A/Etafilcon A/Alphafilcon A | Alphafilcon A/Senofilcon A/Etafilcon A | Etafilcon A/Alphafilcon A/Senofilcon A
Started | 17 | 17 | 16 | 14 | 16 | 16
Completed | 17 | 17 | 15 | 14 | 16 | 16
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Discontinuation | 0 | 0 | 1 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Senofilcon A/Alphafilcon A/Etafilcon A | Alphafilcon A/Etafilcon A/Senofilcon A | Etafilcon A/Senofilcon A/Alphafilcon A | Senofilcon A/Etafilcon A/Alphafilcon A | Alphafilcon A/Senofilcon A/Etafilcon A | Etafilcon A/Alphafilcon A/Senofilcon A
Started | 17 | 17 | 15 | 14 | 16 | 16
Completed | 17 | 17 | 15 | 14 | 16 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Senofilcon A/Alphafilcon A/Etafilcon A | Alphafilcon A/Etafilcon A/Senofilcon A | Etafilcon A/Senofilcon A/Alphafilcon A | Senofilcon A/Etafilcon A/Alphafilcon A | Alphafilcon A/Senofilcon A/Etafilcon A | Etafilcon A/Alphafilcon A/Senofilcon A
Started | 17 | 17 | 15 | 14 | 16 | 16
Completed | 17 | 17 | 14 | 14 | 12 | 14
Not Completed | 0 | 0 | 1 | 0 | 4 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Completed Population: Only participants that completed the study are included (n=88)
Arm/Group | Completed Population
Number analyzed (Participants) | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (5.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Number of eyes with Distance Visual Acuity 20/20 or better
Time Frame: 15-20 minutes
Population: Analysis includes participants who completed the study per protocol (n=88 subjects,176 eyes)
Measure: Number; unit: Eyes with Snellen VA 20/20 or better
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric | Etafilcon A Sphere
Number analyzed (Participants) | 88 | 88 | 88
Eyes with Snellen VA 20/20 or better | 146 | 136 | 37
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Etafilcon A Sphere; Alternative hypothesis was senofilcon A toric was superior to etafilcon A sphere by having more eyes see 20/20; Test type: Superiority or Other; p < 0.0001, Chi-squared

2. Primary Outcome: Patient Reported Vision
Description: A weighted combined score calculated from individual confort-vision related questions asked on a 1-5 scale, 1=most negative resonse to 5=most positive response, was used to derive vision scores. The analysis shows the difference in outcome between test and control. >0=greater vision, <0=lesser vision.
Time Frame: 15-20 minutes
Population: Analysis includes participants who completed the study per protocol (n=88)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric | Etafilcon A Sphere
Number analyzed (Participants) | 88 | 88 | 88
Scores on a scale | 0.2845 (0.098) | 0.1332 (0.098) | -0.4310 (0.097)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Etafilcon A Sphere; Alternative hypothesis was senofilcon A toric was superior to etafilcon A sphere; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.7155, 95% CI [0.3625 to 0.7155], Standard Error of Mean 0.1334 — Mean difference was senofilcon A toric minus etafilcon A sphere

3. Primary Outcome: Lens Orientation Within 5 Degrees
Description: Meaures in what position does the lens sit on the eye at insertion and is measured in degrees of rotation.
Time Frame: 1 minute
Population: Analysis includes participants who completed the study per protocol (n=88 subjects, 176 eyes)
Measure: Number; unit: degrees
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric
Number analyzed (Participants) | 88 | 88
degrees | 142 | 126
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Alphafilcon A Toric; Aletrnative hypothesis was senofilcon A toric was superior to alphafilcon A toric by having more eyes within 5 degrees; Test type: Superiority or Other; p = 0.2161, Chi-squared

4. Primary Outcome: Lens Stability Within 5 Degrees
Description: Measures if the lens changes position on the eye as it is worn and is measured in degrees of rotation.
Time Frame: 1 minute
Population: Analysis includes participants who completed the study per protocol (n=88 subjects, 176 eyes)
Measure: Number; unit: degrees
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric
Number analyzed (Participants) | 88 | 88
degrees | 156 | 140
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Alphafilcon A Toric; Alternative hypothesis was senofilcon A toric was superior to alphafilcon A toric by having more eyes within 5 degrees; Test type: Superiority or Other; p = 0.1328, Chi-squared

5. Primary Outcome: Patient Reported Comfort.
Description: A weighted combined score calculated from individual comfort-related questions asked on a 1-5 scale, 1=most negative response to 5=most positive response, was used to derive comfort outcomes. The analysis shows the difference in outcome between the test and control. >0=comfortable, <0=uncomfortable
Time Frame: 15-20 minutes
Population: Analysis includes participants who completed the study per protocol (n=88)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric | Etafilcon A Sphere
Number analyzed (Participants) | 88 | 88 | 88
Scores on a scale | 0.1425 (0.1034) | -0.3464 (0.1035) | 0.2176 (0.1028)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Alphafilcon A Toric; Alternative hypothesis was senofilcon A toric was superior to alphafilcon A toric; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.4890, 95% CI [0.1529 to 0.4890], Standard Error of Mean 0.1393 — Mean difference was senofilcon A toric minus alphafilcon A toric

6. Primary Outcome: Patient Preference
Description: This outcome measures which lens the subjects preferred to wear.
Time Frame: end of study
Population: Analysis includes participants who completed the study per protocol (n=88)
Measure: Number; unit: Number of participants
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric | Etafilcon A Sphere
Number analyzed (Participants) | 88 | 88 | 88
Number of participants | 62 | 5 | 18
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Etafilcon A Sphere; Alternative hypothesis was senofilcon A toric was superior to etafilcon A sphere; Test type: Superiority or Other; p < 0.0001, Chi-squared

ADVERSE EVENTS:
Arm/Group | Senofilcon A/Alphafilcon A/Etafilcon A | Alphafilcon A/Etafilcon A/Senofilcon A | Etafilcon A/Senofilcon A/Alphafilcon A | Senofilcon A/Etafilcon A/Alphafilcon A | Alphafilcon A/Senofilcon A/Etafilcon A | Etafilcon A/Alphafilcon A/Senofilcon A
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/16 | 0/14 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/16 | 0/14 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.